CLINICAL TRIAL: NCT04924790
Title: The Effect of the COVID-19 Pandemic on Patient Preferences and Decision Making for Obstructive Urinary Stone Interventions
Brief Title: The Effect of the COVID-19 on Patient Preferences and Decision Making for Obstructive Urinary Stone Interventions
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ankara Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Ali Kaan Yildiz, Principal Investigator, Ankara Training and Research Hospital
Other Study IDs: COVIDUS2021
Record Dates: First submitted 2021-06-10; First posted 2021-06-14 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Urinary Stone; Urinary Calculi; Covid19
Keywords: Urinary stone; Obstructive stone; Covid19; Stone surgery
MeSH Terms: conditions — Urinary Calculi; COVID-19 | interventions — Pandemic Preparedness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- COVID-19 Urinary Stone: Patients diagnosed with obstructive urinary stones in the COVID-19 period
  Interventions: Behavioral: COVID-19 Pandemic
- PreCOVID-19 Urinary Stone: Patients diagnosed with obstructive urinary stones in the preCOVID-19 period
  Interventions: Behavioral: COVID-19 Pandemic

INTERVENTIONS:
Behavioral: COVID-19 Pandemic — Comparison of the intervention preferences of patients diagnosed with obstructive urinary stones in the urology clinic and recommended for intervention during and before COVID-19

SUMMARY:
In this study, the investigators aim to evaluate the intervention preferences of patients with obstructive urinary stones who are suitable for operation during the COVID-19 pandemic. The secondary aim is to compare and evaluate the preferences compared to the pre-pandemic period and to gain a perspective on how the decision-making process has changed from the patient's point of view. Thus, by trying to understand how the COVID-19 epidemic affects the treatment choice decisions of patients, the investigators aim to determine how the state of anxiety changes these preferences.

DETAILED DESCRIPTION:
The transformative impact of the COVID-19 pandemic on healthcare use remains an open question. At the onset of the pandemic, policies to limit transmission were adopted, including stay-at-home decisions, social distancing, and postponing elective surgery. Such policies have contributed to reduced emergency room admissions, increased concern about COVID-19, and hospital systems have had to prioritize emergency intervention.

Obstructive urolithiasis is a clinical condition that usually causes severe flank pain and causes emergency admission. It is still unclear how the epidemic impairs the treatment pathways of the obstructive urolithiasis that contributes to the emergency room visit. Treatment options range from observation and medical expulsive therapy to operative interventions such as extracorporeal shock wave lithotripsy, ureteroscopy and percutaneous nephrolithotomy. Patient preference, stone characteristics and comorbidities are of great importance in decision making. However, since obstructive ureteral stones that cannot be resolved spontaneously can cause irreversible renal parenchymal damage and obstructive pyelonephritis in a short time, the option of operation is always prioritized.

Patient perspectives on how COVID-19 is changing healthcare use and decision-making still remain unclear. In our study, the investigators plan to record patient treatment preferences by explaining in detail how and where treatment options will be applied, success and complication rates for patients diagnosed with obstructive urolithiasis and suitable for intervention in the outpatient clinic. In addition, when evaluating patient preferences, the investigators foresee to determine how the COVID-19 pandemic process has changed compared to before. It is planned that our study will have a patient-centered approach with detailed oral and written information in outpatient clinic conditions.

ELIGIBILITY:
Inclusion Criteria:

* Obstructive Urinary Stone

Exclusion Criteria:

* Previous operation for urinary stone
* Presence of bladder stone
* Presence of stent in the ureter
* Previous radiotherapy to the pelvic and abdominal region
* Pregnancy
* Neurological disease

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with obstructive urinary stones in the urology clinic and recommended intervention
Sampling Method: Probability Sample
Enrollment: 158 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-05-01 (Estimated); Study Completion 2022-08-01 (Estimated)

PRIMARY OUTCOMES:
Rates of interventions preferred by patients | 6 months
  Rates of interventions preferred by patients for obstructive urinary stones

CONTACTS AND LOCATIONS:
Overall Officials: Ali Kaan Yildiz, Principal Investigator — Ankara Training and Resarch Hospital
Locations (1):
- Ankara Training and Research Hospital, Ankara, Altindag, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jiang T, Osadchiy V, Weinberger JM, Zheng MH, Owen MH, Leonard SA, Mills JN, Kachroo N, Eleswarapu SV. Impact of the COVID-19 Pandemic on Patient Preferences and Decision Making for Symptomatic Urolithiasis. J Endourol. 2021 Aug;35(8):1250-1256. doi: 10.1089/end.2020.1141. Epub 2021 Mar 4. PMID 33478351
- [Background] Campi R, Tellini R, Grosso AA, Amparore D, Mari A, Viola L, Cocci A, Polverino P, Checcucci E, Alessio P, Fiori C, Minervini A, Carini M, Porpiglia F, Serni S. Deferring Elective Urologic Surgery During the COVID-19 Pandemic: The Patients' Perspective. Urology. 2021 Jan;147:21-26. doi: 10.1016/j.urology.2020.09.015. Epub 2020 Sep 24. PMID 32979378
- [Background] Lee EH, Kim SH, Shin JH, Park SB, Chi BH, Hwang JH. Effects on renal outcome of concomitant acute pyelonephritis, acute kidney injury and obstruction duration in obstructive uropathy by urolithiasis: a retrospective cohort study. BMJ Open. 2019 Nov 3;9(11):e030438. doi: 10.1136/bmjopen-2019-030438. PMID 31685503